CLINICAL TRIAL: NCT03504267
Title: The Influence of Evidence-based Educational Materials and Local Resources in Improving Physical Activity-related Outcomes Among Pregnant Women
Brief Title: Evidence-based Educational Materials and Local Resources for Improving Exercise-related Outcomes During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-225; 5P20GM1034 (Other Grant/Funding Number: NIH NIGMS IDeA Grant)
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy Related; Obesity
Keywords: physical activity; exercise; patient-provider communication
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Health Resources

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Group (Experimental): The PAG (physical activity) group will receive evidence-based educational information as well as a list of local resources for pursuing physical activity.
  Interventions: Other: Physical Activity Education and Resources
- Standard of Care Group (No Intervention): The SOC (standard of care) group will receive no additional information beyond standard-of-care brochures and information

INTERVENTIONS:
Other: Physical Activity Education and Resources — The intervention involves receiving evidence-based educational brochures as well as a list of local facilities where the participant can work out at no-cost to them,
  Arms: Physical Activity Group

SUMMARY:
Despite the well-established benefits of physical activity, only 23% of pregnant women report exercising in accordance with guidelines recommended by the American Congress of Obstetricians and Gynecologists. Further, pregnant women report receiving little or no advice about physical activity during pregnancy from their health care provider; thus, the scientific evidence supporting physical activity during pregnancy does not appear to be translating into the clinic and the community. The goal of this project is to determine if the distribution of evidence-based educational materials and local resources will increase knowledge regarding the benefits of physical activity during pregnancy, patient-provider communication about physical activity during pregnancy, and physical activity levels during pregnancy.

Hypothesis A: Pregnant women who receive evidence-based educational materials and local resources will have increased knowledge regarding the benefits of physical activity during pregnancy.

Hypothesis B: Pregnant women who receive evidence-based educational materials and local resources will have more communication with their health care provider about physical activity.

Hypothesis C: Pregnant women who receive educational information and local resources will report increased physical activity levels.

Hypothesis D: Pregnant women who receive evidence-based educational materials and local resources will have improved pregnancy outcomes including lower gestational weight gain, lower insulin resistance (as determined by their clinical oral glucose tolerance test), and healthier neonatal birthweight.

DETAILED DESCRIPTION:
Physical activity during pregnancy has been shown to be safe and effective in improving maternal and neonatal short and long-term outcomes. Despite all of the benefits, only 23% of all pregnant women report exercising in accordance with guidelines recommended by the American Congress of Obstetricians and Gynecologists. Further, pregnant women report receiving little or no advice about physical activity during pregnancy from their health care provider; thus, the scientific evidence supporting exercise during pregnancy does not appear to be translating into the clinic and the community. With maternal obesity becoming a serious public health concern, the need for awareness and communication about physical activity during pregnancy is more important than ever before. Kentucky-specific data suggests that the incidence of obesity at the first prenatal visit has increased from 7% to 24% over the past 20 years, and local interventions to reduce obesity during pregnancy are limited. Thus, physical activity interventions designed to combat obesity and improve maternal and neonatal health are warranted, specifically in rural Kentucky where rates of obesity and physical inactivity are considerably higher than the national averages. A goal of this project is that it will be the start of a sustainable program that will improve the lives of pregnant women and their neonates in the community. The proposed program can grow beyond the city of Bowling Green, KY, and this model can be adopted across the state of Kentucky. This program will not only educate the population about all of the benefits of physical activity during pregnancy (which is important as a previous study demonstrated that rural communities have perceptions that support myths about exercise during pregnancy), but it will increase physical activity levels among pregnant women. The long-term impact of increased maternal physical activity levels in the city, state, and nation is substantial as many studies have shown that physical activity during pregnancy has a long-term impact of maternal and neonatal health outcomes.

Because Kentucky is one of the most obese states in America, it is important local interventions are designed to reduce obesity in future generations in order to stop the vicious cycle of obesity. If the program succeeds and grows, it has the potential to improve the overall health of the city of Bowling Green (and beyond) for years to come. Although obesity is a multifaceted issue, and much larger steps need to be taken at the national level to combat it, programs such as this are a small step in the right direction. Intervening as early as possible (neonatal level) is an important opportunity to improve health in future generations. Previous studies have demonstrated that antenatal lifestyle advice improves maternal physical activity during pregnancy, and that information regarding risks and benefits of exercise during pregnancy can be a source of exercise motivation for pregnant women. In addition,this study design removes common barriers to participating in physical activity during pregnancy by providing a number of medically-supervised exercise options (one of which offers childcare, one of which can be done without leaving the home, and many of which have safe and comfortable options for pregnant women), all at no cost to the pregnant women.

The goals of Specific Aim 2 are to increase patient awareness about the benefits of physical activity during pregnancy, increase patient-provider communication about physical activity during pregnancy, and increase physical activity levels during pregnancy in rural Kentucky through the use of evidence-based educational materials and local resources.

The study team hypothesizes that providing pregnant women with evidence-based educational materials and a selection of local resources will increase knowledge about the benefits and risks of physical activity, increase patient-provider communication about physical activity, and increase physical activity levels during pregnancy. If physical activity levels are increased, this study may also help to improve maternal and neonatal outcomes. This study may help pregnant women gain less weight during pregnancy, and thus, combat maternal obesity in the years following pregnancy.In addition, this study may contribute to healthier offspring as physical activity during pregnancy has been shown to reduce offspring birth weight and body fat percentage into childhood.

All participants (N=80) will be recruited from Graves Gilbert Obstetrics, a rural healthcare clinic, between 8 and 12 weeks gestation. Once consented to participate, all women will take baseline surveys between 8 and 12 weeks gestation. Surveys will be taken before or after their prenatal appointment at Graves-Gilbert. If this is not feasible for the participant, surveys can be taken home and mailed back to the study team upon completion. Baseline surveys will assess knowledge, beliefs, and motivation to be physically active during the index pregnancy. In addition, all women will be asked to report physical activity levels during their pregnancy. In addition to surveys about physical activity during pregnancy, all participants will also receive a Xaomi Mi Band, a wrist-worn physical activity monitor that calculates steps and kilocalories expended per day for 30 days at a time. If possible, participants will be asked to sync the device with their smart phone and text the study team information regarding their steps and energy expenditure. If this is not feasible, the study team will meet them once a month at their clinic appointment and sync the data directly to a portable laptop device. After baseline surveys are complete, each participant will be randomized to the physical activity group (PAG) or the standard of care group (SOC). The PAG will receive evidence-based educational information as well as a list of local resources for pursuing physical activity. Local resources will be provided to the pregnant women in the study at no charge, thus, financial constraints will not be a barrier to physical activity during pregnancy for women in the present study. SOC will receive no additional information beyond standard-of-care brochures and information. At 32-34 weeks gestation, all women will be surveyed once again regarding knowledge and beliefs, motivation, and physical activity levels during their pregnancy. The Dietary History Questionnaire II will also be administered in order to control for dietary differences between groups that could contribute to outcomes being assessed. In addition to the baseline surveys, all women will be surveyed about patient-provider communication regarding physical activity during their pregnancy. Outcomes will be compared between PAG and SOC groups. Prenatal charts will be obtained after infant delivery. Additional maternal and neonatal outcomes will be examined to determine the effect of the intervention on outcomes (i.e. gestational weight gain, postpartum weight retention, oral glucose tolerance test results, neonatal birth weight).

The evidence-based educational materials are adopted from previous research that demonstrated educational materials motivate pregnant women to exercise as well as alter their beliefs about physical activity during pregnancy The evidence-based brochure has been designed and made culturally appropriate. Surveys were designed using constructs of the Theory of Planned Behavior (knowledge and beliefs) and the Protection Motivation Theory and Health Action Process Approach (motivation).

Statistical Procedures Repeated measures ANOVAs will be used to compare scores on the Exercise Belief's Questionnaire I (agree/disagree) and physical activity levels (PPAQ, Mi Band data) between the two groups before and after the intervention. Motivation outcomes will be assessed by identifying recurring themes in relation to the Protection Motivation Theory and Health Action Process Approach and comparing responses between groups. Recurrent themes will be identified regarding the Exercise Beliefs Questionnaire II, and improvement will be based on the number of correct responses for each question before and after the intervention. Patient-provider communication frequency and topic will be compared between the groups using chi-square tests. All tests will be two-sided with a p-value <0.05 denoting statistical significance. All data analyses will be conducted using IBM SPSS Statistics, Version 22 (Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44
* Confirmed singleton viable pregnancy
* English-Speaking

Exclusion criteria:

* Multiple gestation pregnancy
* Inability to provide voluntary informed consent
* Any medical condition (pregnancy-related or not) that would preclude exercise

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge regarding physical activity during pregnancy | Change in knowledge from baseline (8-12 weeks) to late gestation (32-34 weeks)
  Validated survey tools from previous studies (and tested in a separate cohort of local women)
Change in physical activity levels | Change in steps per day from baseline (8-12 weeks) to late gestation (32-34 weeks)
  Mi-Band devices will be worn on the wrist for one week at each time point

SECONDARY OUTCOMES:
Patient-provider communication | This will be assessed at the end of pregnancy (32-34 weeks) by both the patient and the provider
  Previously used surveys developed by the PI
Gestational weight gain | Change in body weight from pre-pregnancy (self-reported at enrollment (kg) to the very end of pregnancy(~40 weeks gestation) (kg))
  Total weight gained during pregnancy
Insulin resistance | 28 weeks gestation
  Oral glucose tolerance test results
Infant birth weight | At study completion, ~ 40 weeks gestation
  Self-reported weight of the baby at the time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Tinius, PhD, Principal Investigator — Western Kentucky University
Locations (1):
- Graves Gilbert Obstetric Clinic, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No